CLINICAL TRIAL: NCT05515003
Title: Evaluation of the Effect of Patient Education on the Management of Fatigue and Quality of Life in Individuals With Inflammatory Bowel Disease
Brief Title: The Effect of Patient Education on Fatigue and Quality of Life in Inflammatory Bowel Disease
Acronym: IBD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Collaborators: Eskisehir Osmangazi University (Other)
Responsible Party: Principal Investigator, Zeliha Tülek, RN,Assoc Prof, Istanbul University - Cerrahpasa
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Fatigue
Record Dates: First submitted 2022-08-23; First posted 2022-08-25 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Inflammatory Bowel Diseases
Keywords: Fatigue; Quality of life
MeSH Terms: conditions — Inflammatory Bowel Diseases; Fatigue

STUDY DESIGN:
Intervention Model Description: Nonrandomized Control Group, Pretest-Posttest Design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Education group (Experimental): Individualized patient education
  Interventions: Other: Individualized patient education
- Control group (No Intervention): No training will be provided

INTERVENTIONS:
Other: Individualized patient education — In the intervention group, patients will undergo a single, personalized education session led by the researcher, lasting 30 to 60 minutes. Identified knowledge gaps will be addressed through focused education, followed by interactive question-and-answer sessions covering fatigue, diarrhea/constipation, abdominal pain, mental health, nutrition, exercise, and sleep.
  Follow-up calls will be conducted in the 1st, 2nd, and 3rd weeks post-education to monitor patient progress. Each call will assess general health status, symptom severity, and changes in bowel habits. Patients will be encouraged to review educational materials and ask questions, with appointment reminders provided during the 3rd week. These calls will each last approximately 10-15 minutes.
  One month later, follow-up interviews will evaluate the education's impact using updated data collection tools, ensuring a thorough assessment of its effect on patient outcomes.
  Arms: Education group

SUMMARY:
Introduction: Fatigue is a serious symptom that is seen in a significant portion of IBD patients and negatively affects the patient's quality of life. The aim of this study is to evaluate the effect of patient education on the management of fatigue, which is common in inflammatory bowel diseases.

Material and methods: This study will be planned with nonrandomized control group, pretest-posttest design. It is planned that the sample group will consist of at least 84 patients, 42 of which are in the intervention group and 42 in the control group. The patients in the intervention group will be evaluated in terms of fatigue and factors that may affect it, and an individualized education program will be offered according to the needs of the patient.For the patients in the control group, only the scales used in data collection will be filled, and no education will be planned. One month after the first interviews, both groups will fill in the scales again.

DETAILED DESCRIPTION:
The aim of this study is to evaluate the effect of patient education on the management of fatigue, which is common in inflammatory bowel diseases.This study will be conducted in IBD outpatient clinic in Eskisehir Osmangazi University Hospital. This study will be planned with a nonrandomized control group, pretest-posttest design. Patients who meet the criteria will be assigned to the intervention or control group. It is planned that the sample group will consist of at least 84 patients, 42 of which are in the intervention group and 42 in the control group. The patients in the intervention group will be evaluated in terms of fatigue and factors that may affect it, and an individualized education program will be offered according to the needs of the patient. All patients will be assessed at baseline by use of following tools: Patient Information Form, Crohn's Disease Harvey-Bradshaw Activity Index (HBI), Simple Colitis Clinical Activity Index (SCCAI), Inflammatory Bowel Diseases Fatigue (IBD-F) Scale, Inflammatory Bowel Diseases Quality of Life Assessment Questionnaire. Patients in the intervention group will be applied one-session individualized patient education by the researcher. The control group will be applied usual care. Two groups will be compared at baseline and at the 1st month after the intervention with the same scales

ELIGIBILITY:
Inclusion Criteria:

* Disease in remission
* Diagnosis of inflammatory bowel disease with endoscopic procedures
* Being over 18 years old,
* Patient's volunteering to participate in the research

Exclusion Criteria:

* Having a psychiatric illness,
* Having a diagnosis of chronic fatigue syndrome,
* Difficulty in communicating (speech, perception, understanding problem),
* Having an advanced chronic disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2023-09-27 (Actual)

PRIMARY OUTCOMES:
Change in the Inflammatory Bowel Disease Fatigue Patient Self-Assessment Scale scores | At the baseline, 1st month after the intervention
  Fatigue will be assessed with the Inflammatory Bowel Disease Fatigue Patient Self-Assessment Scale. The scale was developed to diagnose fatigue or to monitor the level of fatigue over time. The scale consists of three sections. A score of 0-20 can be obtained from Section 1. A score of 0 means no fatigue. Therefore, there is no need to complete sections 2 and 3. A score of 1-10 means mild to moderate fatigue, and a score of 11-20 means severe fatigue. A score between 0--120 can be obtained from Section 2. A score of 0 indicates that fatigue does not affect daily activities, a score of 1-60 indicates that it affects it moderately, and a score of 61-120 indicates that it affects it severely. Section 3 is not scored. Higher scores indicate a higher level of fatigue (Section I) or the severity of the impact of fatigue on an individual's life (Section II).

SECONDARY OUTCOMES:
Change in the Inflammatory Bowel Diseases Quality of Life Scale scores | At the baseline, 1st month after the intervention
  Quality of life will be assessed with the Inflammatory Bowel Disease Quality of Life Questionnaire. Quality of life will be assessed with the Inflammatory Bowel Disease Quality of Life Questionnaire. Scores ranging from 36 to 252 can be obtained from the questionnaire. As the score obtained from the scale increases, the quality of life of the patients also increases.

CONTACTS AND LOCATIONS:
Overall Officials: ZELIHA TULEK, Assoc.Prof., Study Director — Istanbul University-Cerrahpasa, Florence Nightingale Faculty of Nursing
Locations (1):
- Eskisehir Osmangazi University, Eskişehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tiles-Sar N, Neuser J, de Sordi D, Baltes A, Preiss JC, Moser G, Timmer A. Psychological interventions for treatment of inflammatory bowel disease. Cochrane Database Syst Rev. 2025 Apr 17;4(4):CD006913. doi: 10.1002/14651858.CD006913.pub3. PMID 40243391